CLINICAL TRIAL: NCT00000753
Title: A Phase I Concentration-Targeted Multidose Study of Atevirdine Mesylate ( U-87201E ), AZT, and ddI or ddC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Upjohn (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 187; 11162 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — atevirdine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Atevirdine mesylate
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To determine the safety, toxicity, pharmacokinetic profile, and antiretroviral activity of atevirdine mesylate ( U-87201E ) in HIV-infected patients. Per 06/04/93 amendment, to also evaluate the interactive effects of didanosine ( ddI ) or zalcitabine ( dideoxycytidine; ddC ) with zidovudine ( AZT ) on the pharmacokinetics of U-87201E and to assess the effects of the triple combination therapies on immunologic and virologic parameters.

Since the use of non-nucleoside reverse transcriptase inhibitors such as U-87201E has been associated with the rapid development of resistant HIV isolates, an initial evaluation of this drug in patients was made in combination with AZT. Because of the inability to detect resistance after 6 weeks of combined AZT/U-87201E therapy, this protocol will initially investigate U-87201E administered alone and then investigate the effect of this drug with AZT and ddI or ddC.

DETAILED DESCRIPTION:
Since the use of non-nucleoside reverse transcriptase inhibitors such as U-87201E has been associated with the rapid development of resistant HIV isolates, an initial evaluation of this drug in patients was made in combination with AZT. Because of the inability to detect resistance after 6 weeks of combined AZT/U-87201E therapy, this protocol will initially investigate U-87201E administered alone and then investigate the effect of this drug with AZT and ddI or ddC.

Ten patients are treated at each of three targeted concentration ranges of U-87201E. Patients in the second cohort are enrolled immediately after patients in the first cohort are accrued; patients in the third cohort are enrolled when 5 of 10 patients in the second cohort have tolerated that dose for at least 4 weeks. The MTD will be the dose below that which produces dose-limiting grade 3 or 4 toxicity in five out of 10 patients. At least two women and five antiretroviral naive patients must be enrolled in each dose concentration range. Patients receive at least 8 weeks of monotherapy with U-87201E, with possible extension to at least 24 weeks with the same dose of U-87201E alone or in combination with zidovudine plus either ddI or ddC. Patients are followed weekly for at least 8 weeks and, if applicable, at weeks 10, 12, 16, 20, and 24 and monthly thereafter, up to 1 month following the last dose. Patients on combination therapy will have an indwelling venous catheter inserted for the first 2 days of combination therapy. Per 10/15/93 amendment, if no MTD is established with the first three cohorts, then 10 additional patients will be enrolled at a fourth concentration.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis with pentamidine, TMP/SMX, or dapsone (if appropriate).
* Clotrimazole troches or nystatin oral suspension for oral candidiasis.
* Acyclovir (up to 1000 mg/day) for herpes lesions.
* Supportive care as deemed necessary for toxicities .

Patients must have:

* HIV infection.
* CD4 count <= 500 cells/mm3.
* No active opportunistic infections.
* Consent of parent, guardian, or person with power of attorney, if less than 18 years of age.

NOTE:

* Participation of women in the study is encouraged.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Acute medical problems, including opportunistic infections (e.g., active cryptococcosis, Pneumocystis carinii, herpes zoster, histoplasmosis, and CMV) or nonopportunistic diseases (e.g., liver or renal disease or lymphoma).
* Current diagnosis of malignancy for which systemic therapy would be required during the study.
* Active gastrointestinal disorders.

Concurrent Medication:

Excluded:

* Investigational drugs.
* Systemic therapy for malignancy.
* Phenobarbital, phenytoin, ketoconazole, rifampin, rifabutin, cimetidine, beta blockers, chronic antacids, antiarrhythmic agents, or other medications known to affect cardiac conduction or seizure threshold.

Patients with the following prior conditions are excluded:

* History of any cardiovascular disease, including conduction disturbances, arrhythmias or atherosclerotic heart disease.
* History of CNS disease such as seizure disorder, AIDS Dementia Complex, progressive multifocal leukoencephalopathy, or any other active neurological disorder.
* History of chronic gastrointestinal disorders such as chronic diarrhea (> 4 weeks duration).

Prior Medication:

Excluded:

* Antiretroviral or immunomodulator agents (such as AZT, ddI, ddC, interferon, etc.) within 15 days prior to study entry.
* Cytotoxic chemotherapy within 1 month prior to study entry.
* Prior U-87201E or other non-nucleoside reverse transcriptase inhibitors (i.e., nevirapine, TIBO, L697,661).

Present use of alcohol or illicit drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reichman R, Study Chair
Locations (6):
- United States (6):
  - USC CRS, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio

REFERENCES:
- [Background] Demeter LM, Meehan PM, Morse G, Fischl MA, Para M, Powderly W, Leedom J, Holden-Wiltse J, Greisberger C, Wood K, Timpone J Jr, Wathen LK, Nevin T, Resnick L, Batts DH, Reichman RC. Phase I study of atevirdine mesylate (U-87201E) monotherapy in HIV-1-infected patients. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Oct 1;19(2):135-44. doi: 10.1097/00042560-199810010-00006. PMID 9768622
- [Background] Morse GD, Reichman RC, Fischl MA, Para M, Leedom J, Powderly W, Demeter LM, Resnick L, Bassiakos Y, Timpone J, Cox S, Batts D. Concentration-targeted phase I trials of atevirdine mesylate in patients with HIV infection: dosage requirements and pharmacokinetic studies. The ACTG 187 and 199 study teams. Antiviral Res. 2000 Jan;45(1):47-58. doi: 10.1016/s0166-3542(99)00073-x. PMID 10774589